CLINICAL TRIAL: NCT04011384
Title: A Randomized Trial of Web-based Behavioral Economic Interventions to Promote Healthy Food Choices Among Food Pantry Clients
Brief Title: A Trial of Behavioral Economic Interventions Among Food Pantry Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Massachusetts General Hospital (Other); University of Connecticut (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christina Roberto, Assistant Professor of Medical Ethics & Health Policy, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPCC 06022; R01CA229502 (NIH); 829702 (Other: IRB)
Record Dates: First submitted 2019-07-05; First posted 2019-07-08 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Food Preferences
Keywords: Food Assistance; Economics, Behavioral; Food Labeling; Diet Records; Biomarkers
MeSH Terms: conditions — Food Preferences; Behavior

STUDY DESIGN:
Intervention Model Description: The researchers will recruit 500 regular food pantry clients to participate in a randomized-controlled trial that involves visiting the food pantry and selecting food using the web-based ordering system, having physical measurements collected by study staff, completing food frequency questionnaires, completing a health survey, and getting a blood draw to measure fruit and vegetable intake and health outcomes from biomarkers. Participants will be randomized to 1 of 2 conditions: 1) control group (usual care); or 2) behavioral economic intervention group.
Who Masked: Investigator
Masking Description: The research team will create the randomization list and a research assistant will assign the participant to the correct online platform condition, but the investigators and data analysts will remain blind to group assignment. This study will contain two parallel groups. Although participants will not initially be aware of the other study condition, they will not be blinded to study condition because those in the intervention condition will be viewing the altered ordering platform as they shop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in this arm will view the typical web-based ordering system platform (usual care group).
- Behavioral Economic Intervention Group (Experimental): Participants in this arm will be exposed to the web-based ordering system with multiple behavioral economic interventions applied, including healthy food shopping cart defaults, healthy placement choice architecture, traffic light nutrition labels, social norms messaging, and healthy swaps.
  Interventions: Behavioral: Behavioral economic intervention of online purchasing at a food pantry

INTERVENTIONS:
Behavioral: Behavioral economic intervention of online purchasing at a food pantry — This intervention includes multiple behavioral economic interventions, healthy food shopping cart defaults, healthy placement choice architecture, traffic light nutrition labels, social norms messaging, and healthy swaps.
  Arms: Behavioral Economic Intervention Group

SUMMARY:
Obesity, unhealthy dietary habits, and food insecurity are major public health concerns, especially affecting individuals living in poverty. Food pantries, which provide free food to those in need, are increasingly interested in promoting healthy choices, but few rigorous studies have tested healthy eating interventions in food pantry settings. The overall objective of this proposal is to conduct a randomized-controlled trial among 500 regular food pantry clients to compare the influence of a behavioral economic intervention to promote healthier food choices delivered via a web-based ordering platform to usual care (control group).

DETAILED DESCRIPTION:
The primary objective of this proposal is to evaluate the influence of a web-based behavioral economic intervention compared to a control group on the following outcomes among food pantry clients: 1) Nutritional quality of food chosen at the pantry using food transaction data; 2) Fruit and vegetable intake measured by biomarkers and food frequency questionnaires; 3) Objectively measured biomarkers of health. The web-based behavioral economic intervention will include the following modifications to the online shopping platform: 1) Healthy food shopping cart defaults, 2) healthy placement choice architecture, 3) traffic light nutrition labels, 4) social norms messaging, and 5) healthy swaps. Food transaction data will be collected from the online system at baseline and then continuously for the remaining 3 months of the study (participants typically shop monthly). Surveys and objective biomarkers will be collected at baseline and three-months.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* primary grocery shopper for the family
* a regular in-person client at the food pantry (i.e., shops at pantry ≥ 1 per month)
* able to use the web-based touchscreen ordering system
* able to use a blood pressure cuff and scale provided to them for taking blood pressure and weight
* able to come outside their home for 5 minutes for the Veggie Meter measurement

Exclusion Criteria:

* <18 years old
* not the primary grocery shopper for the family
* not a regular client at the food pantry (i.e., shops at pantry < 1 per month)
* not able to use the web-based touchscreen ordering system
* not able to use a blood pressure cuff and scale provided to them for taking blood pressure and weight
* not able to come outside their home for 5 minutes for the Veggie Meter measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were clients at a food pantry and were recruited either in-person at the pantry or by phone (after March 2020 due to the Covid-19 pandemic). Recruitment ran from July 2019 to September 2022. 70% of participants were recruited before the pandemic.
Pre-assignment Details: Due to the Covid-19 pandemic, we lost 47 participants who were consented (before March 2020), but had not yet completed their baseline appointment. 3 others were accidentally enrolled, but did not meet our enrollment criteria and were excluded before baseline. Finally 1 was excluded because they were not randomized to a condition.
Period: Overall Study
Arm/Group | Control Group | Behavioral Economic Intervention Group
Started | 111 | 124
Completed | 109 | 124
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Behavioral Economic Intervention Group | Total
Number analyzed (Participants) | 109 | 124 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 66 (15) | 66 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 91 | 156
  Male | 44 | 33 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 105 | 121 | 226
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 88 | 109 | 197
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 4 | 0 | 4
Language [Count of Participants; unit: Participants]
  English | 50 | 55 | 105
  Russian | 56 | 66 | 122
  Other language | 3 | 3 | 6
Education [Count of Participants; unit: Participants]
  Less than high school | 5 | 6 | 11
  High school degree or equivalent | 30 | 29 | 59
  Some college or associates | 24 | 33 | 57
  College or above | 49 | 53 | 102
  Unknown | 1 | 3 | 4
Children at home [Count of Participants; unit: Participants]
  No children at home | 87 | 105 | 192
  1 or more children at home | 19 | 17 | 36
  Unknown | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Monthly Change in Number of Units of Healthier Foods
Description: Average monthly change from baseline across 3 months of participation, in number of units of healthier foods (labeled with a green traffic light) purchased per shopping trip using the food pantry's definition of a unit.
Time Frame: Collected from the online system at baseline and then each month for the remaining 3 months of participation.
Population: Some participants were missing order data -- especially near March 2020 at the start of the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: units of healthy food
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 99 | 107
units of healthy food | -1.32 (7.77) | 0.53 (5.54)

2. Primary Outcome: Mean Monthly Change in Number of Units of Less Healthy Foods
Description: Average monthly change from baseline across 3 months of participation, in number of units of less healthy foods (labeled with a red or yellow traffic light) purchased per shopping trip using the food pantry's definition of a unit.
Time Frame: Collected from the online system at baseline and then each month for the remaining 3 months of participation.
Population: Some participants were missing order data -- especially near March 2020 at the start of the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: units of less healthy food
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 99 | 107
units of less healthy food | 0.20 (3.67) | -0.04 (2.68)

3. Secondary Outcome: Mean Monthly Change in Calories From Healthier Foods Per Shopping Trip
Description: Average monthly change from baseline across 3 months of participation, in number of calories from healthier foods per shopping trip.
Time Frame: Collected from the online system at baseline and then each month for the remaining 3 months of participation.
Population: Some participants were missing order data -- especially near March 2020 at the start of the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: calories from healthy food
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 99 | 107
calories from healthy food | -124 (694) | 31 (581)

4. Secondary Outcome: Mean Monthly Change in Calories From Less Healthy Foods Per Shopping Trip
Description: Average monthly change from baseline across 3 months of participation, in number of calories from less healthy foods per shopping trip.
Time Frame: Collected from the online system at baseline and then each month for the remaining 3 months of participation.
Population: Some participants were missing order data -- especially near March 2020 at the start of the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: calories from less healthy food
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 99 | 107
calories from less healthy food | 29 (545) | 14 (472)

5. Secondary Outcome: Self-reported Change in Fruit and Vegetable Intake
Description: Change from baseline in fruit and vegetable intake as measured by the National Cancer Institute (NCI)'s fruit and vegetable module of the Dietary Screener Questionnaire in the National Health and Nutrition Examination Survey (NHANES). Scores estimate average daily cup equivalents of total fruit and vegetable servings.
Time Frame: Assessed at baseline and 3 months.
Population: Some participants were missing survey data -- especially near March 2020 at the start of the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: cup equivalents/day
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 97 | 109
cup equivalents/day | -0.01 (1.25) | 0.08 (1.32)

6. Secondary Outcome: Biomarker Change in Fruit and Vegetable Intake
Description: Change from baseline in carotenoid levels (scores range 0-800) as measured by the VeggieMeter®. The VeggieMeter® is a spectroscopy-based skin carotenoid measurement device, created by Longevity Link Corporation in 2015. It uses pressure-mediated reflection spectroscopy (RS) to detect and quantify skin carotenoids as a proxy for fruit and vegetable intake in humans. Validation studies show VeggieMeter scores to be highly correlated with blood serum measures of carotenoids (R=.81). Higher units represent a higher concentration of carotenoids in the skin.
Time Frame: Assessed at baseline and 3 months.
Population: Many participants were unable to complete the 2nd in-person data collection due to Covid-19
Measure: Mean (Standard Deviation); unit: skin carotenoid score
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 53 | 60
skin carotenoid score | 11 (113) | 4 (113)

7. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline in BMI (weight in kg / height in meters^2)
Time Frame: Assessed at baseline and 3 months.
Population: Several participants were not able to do the follow-up in-person measures due to the Covid-19 pandemic
Measure: Mean (Standard Deviation); unit: kilograms per square meter
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 66 | 69
kilograms per square meter | -0.11 (1.48) | -0.12 (1.48)

8. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change from baseline in systolic blood pressure (indicator of heart health)
Time Frame: Assessed at baseline and 3 months.
Population: Several participants were not able to complete the follow-up in-person appointments due to the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 66 | 69
mmHg | 5.3 (16.3) | 0.1 (16.5)

9. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change from baseline in diastolic blood pressure (indicator of heart health)
Time Frame: Assessed at baseline and 3 months.
Population: Several participants were not able to make it to their follow-up in-person appointment due to the Covid-19 pandemic.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Behavioral Economic Intervention Group
Number analyzed (Participants) | 66 | 69
mmHg | 2.5 (11.0) | -0.3 (9.0)

ADVERSE EVENTS:
Time Frame: 4 months, each participant was assessed from baseline through the 3 months of the study
Arm/Group | Control Group | Behavioral Economic Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/124
Other Adverse Events (participants affected / at risk) | 0/109 | 0/124

LIMITATIONS AND CAVEATS:
Recruiting and assessing measurements (height, weight, blood pressure, and carotenoid levels) in person were limited by the onset of the Covid-19 pandemic in the middle of the study. In addition, monthly food pantry use was certainly impacted by the pandemic as well.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT04011384/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT04011384/ICF_002.pdf